CLINICAL TRIAL: NCT04472806
Title: A Multicenter, Single-arm, Open, Phase II Clinical Study on the Efficacy and Safety of Toripalimab(JS001) After Chemotherapy in Combination With Endostar in Patients With Unresectable Locally Advanced or Metastatic Mucosal Melanoma
Brief Title: Maintenance Treatment of Toripalimab(JS001) in Patients With Unresectable Locally Advanced or Metastatic Mucosal Melanoma
Acronym: MTAM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Fujian Cancer Hospital (Other Government); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLuo
Record Dates: First submitted 2020-07-09; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Mucosal Melanoma
MeSH Terms: interventions — toripalimab; Drug Therapy; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chemotherapy+Endostar+Toripalimab(JS001) (Experimental)
  Interventions: Drug: Toripalimab; Drug: chemotherapy in combination with Endostar

INTERVENTIONS:
Drug: Toripalimab — Toripalimab, humanized anti-PD-1 monoclonal antibody is a programmed death-1 (PD-1) immune checkpoint inhibitor antibody, which selectively interferes with the combination of PD-1 with its ligands, PD-L1 and PD-L2, resulting in the activation of lymphocytes and elimination of malignancy theoretically.
  Toripalimab treatment after chemotherapy in combination with Endostar, 240 mg, Q3W, up to 2 years.
  Other Names: JS001
Drug: chemotherapy in combination with Endostar — chemotherapy+ Endostar

SUMMARY:
This study is a multicenter, single-arm, open, phase Ⅱ clinical study to evaluate the safety and efficacy of Toripalimab(JS001) monoclonal injection after chemotherapy in combination with Endostar for Locally Advanced or Metastatic Mucosal Melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, male or female；
2. Histopathologically confirmed and diagnosed as mucosal melanoma;
3. ECOG score 0 or 1;
4. Life expectancy of at least 12 weeks；
5. SD/PR/CR after chemotherapy in combination with Endostar;
6. No contraindications, having adequate organ and marrow function；
7. Use of highly-effective contraceptive methods during the whole study for men of reproduction ability or women of childbearing potential (e.g. oral contraceptives, intrauterine contraceptive device, abstinence of sexual intercourse or barrier contraception in combination with spermatocide), and continuation of contraception for 12 months after the end of treatment；
8. The subject is voluntary to participate in the study, sign the informed consent form, with good compliance and willingness to cooperate with follow-up.

Exclusion Criteria:

1. Previously treated with anti-PD-1, anti-PD-L1, anti-PD-L2;
2. Known allergy to recombinant humanized anti-PD-1 monoclonal antibody drug and its components;
3. Skin melanoma, eye melanoma, melanoma with unknown primary foci;
4. Symptomatic brain or meningeal metastases, unless the patient has been treated for > 6 months, the imaging results are negative within 4 weeks before entering the study, and the clinical symptoms associated with the tumor are stable at the time of entering the study;
5. Female patients who are pregnant or lactating, or of childbearing potential but not using appropriate contraceptive measures;
6. Currently having serious and uncontrolled acute infection; or suppurative infection and chronic infection with prolonged wound healing;
7. Having serious heart disorder, including cardiac failure congestive, uncontrollable high-risk arrhythmia, unstable angina pectoris, infarct myocardial, severe cardiac valve disease and refractory hypertension;
8. Having neurological, mental disease or mental disorder that can not be easily controlled, poor compliance, inability to cooperate and narrate therapeutic response;
9. Patients with other malignant tumors at the same time;
10. Patients participated in other clinical trials at the same time;
11. Positive HIV; positive HCV; positive HBsAg or HBcAb whilst positive HBV DNA copies detected (limit of quantitation 500 IU/mL);
12. Active autoimmune diseases requiring systemic treatment in the past two years (e.g., use of disease-regulating drug, corticosteroid or immunosuppressant), relevant replacement therapy is allowed (e.g., thyroxine, insulin or physiological corticosteroid replacement therapy for renal or pituitary insufficiency);
13. Having received live vaccine within 4 weeks prior to the start of treatment;
14. Other severe, acute or chronic medical diseases or mental diseases or abnormalities in laboratory examination possibly increasing the relevant risk in study participation or possibly interfering the interpretation of study results as judged by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival, PFS | Approximately 1 years
  PFS is defined as the time from the date of first treatment to the first occurrence of disease progression or death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate, ORR | Approximately 2 years
  ORR is defined as the proportion of patients with a complete response (CR) or partial response (PR) on two consecutive occasions >= 4 weeks apart, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1).
Overall Survival, OS | Approximately 2 years
  OS is defined as the time from the date of first treatment to death from any cause.
Incidence of AEs/SAEs | Approximately 2 years
  Percentage of Participants With Adverse Events/Severe Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Zhiguo Luo, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided